CLINICAL TRIAL: NCT02419859
Title: A Prospective, Single Center Study to Assess the Performance, Safety, and Patient Reported Outcomes of Insulin Delivery With PaQ® in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess Insulin Delivery With PaQ® in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CeQur Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQR14002
Record Dates: First submitted 2015-03-24; First posted 2015-04-17 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Insulin; Continuous subcutaneous insulin infusion (CSII); Insulin pumps
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Insulin Resistance | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PaQ® Insulin Delivery Device (Experimental): The intervention is continuous subcutaneous U 100 Insulin, Asp(B28)-rapid-acting insulin, at a constant basal rate of either 20, 24, 32, 40 or 50 U per day over 3 days and and bolus insulin as needed at meals in 2 U increments.
  Interventions: Device: PaQ® Insulin Delivery Device; Drug: Insulin, Asp(B28)-

INTERVENTIONS:
Device: PaQ® Insulin Delivery Device — PaQ is a 3 day insulin delivery device which delivers U 100 rapid-acting insulin. Provides basal insulin at preset basal doses and bolus insulin (in 2 unit increments) with a push of a button.
Drug: Insulin, Asp(B28)- — a fast-acting analog of human insulin
  Other Names: NovoRapid

SUMMARY:
The purpose of the study is to obtain an assessment (efficacy, safety, and patient reported outcomes) of basal bolus insulin delivery with PaQ in insulin-using patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This is a prospective, single center, open-label, uncontrolled study to assess the efficacy, safety, and patient reported outcomes of insulin delivery with PaQ® in patients with type 2 diabetes mellitus (T2DM) who are currently receiving basal/bolus insulin therapy with or without oral anti-diabetic drugs (OADs) for glycemic control. The patient's participation in the study is comprised of three phases: screening/baseline evaluation, transition to PaQ use and optimization, and PaQ treatment period. The use of these phases will allow an orderly transition to PaQ treatment as well as a reliable construct from which to interpret the final data.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age;
* Has a clinical diagnosis of T2DM, as determined by clinical history and medication usage;
* Has an A1C ≥ 7.0% and ≤ 11.0%;
* Is treated with basal-bolus insulin therapy (at least 2 injections per day) with or without OADs, and/or GLP-1 agonist for at least 3 months and has not had a change (addition or discontinuation of existing drug or change in dose) in their OADs for the last 8 weeks, (See Section 7.4 for definition of baseline basal bolus therapy);
* Determined by the investigator that insulin requirements to achieve glycemic targets can be met by the insulin capacity of the PaQ device;
* If on concomitant metformin, has serum creatinine <1.5 mg/dL (male) or <1.4 mg/dL (female);
* If female, and of child-bearing potential, has a negative urine pregnancy test at screening and must be using adequate means of contraception as determined by the Investigator;
* Is clinically euthyroid as judged by the Investigator;
* Is able to understand and sign the required study documents and comply with the CIP requirements;
* Is deemed capable by the Investigator to perform the requirements of the CIP, including use of PaQ, frequent self-monitoring of blood glucose.

Exclusion Criteria:

* Is poorly compliant with the currently prescribed diabetes regimen, as determined by the Investigator;
* Is poorly compliant with prescribed self-monitoring of blood glucose, as determined by the Investigator;
* Is currently taking or has taken sulfonylureas within the last 2 months;
* Has a BMI greater than 40 kg/m2;
* Has experienced recurrent severe hypoglycemia (> 2 episodes) requiring assistance during the past 6 months;
* Has existing dermal irritation/inflammation over the abdominal area that may interfere with use of PaQ, as determined by the Investigator;
* Has known clinically significant hypersensitivity to skin adhesives;
* Is female and if of child-bearing potential, is pregnant, lactating, or planning to become pregnant;
* Is currently being treated with or expected to require or undergo treatment with systemic steroids by oral, intravenous, or intramuscular route (inhaled with low systemic exposure is permitted);
* Currently abuses drugs or alcohol or has a history of abuse that in the Investigator's opinion would cause the individual to be non-compliant;
* Has received any investigational drug within 1 month;
* Has donated blood within 30 days;
* Has any significant medical condition (including current or past history of cardiovascular disease), laboratory findings, or medical history that in the Investigator's opinion may affect successful completion of the study and/or personal well-being;
* Is an immediate family member (spouse, parent, child, or sibling) of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin A1C (HbA1c) (obtained from venous blood) | Change from Baseline at 12 weeks

SECONDARY OUTCOMES:
Glycosylated hemoglobin A1C (HbA1c) (obtained from venous blood) | Change from Baseline at 8 weeks
Fasting plasma glucose | Change from Baseline at 12 weeks
7-point blood glucose profiles | Change from Baseline at 12 weeks
Total daily dose of insulin | Change from Baseline at 12 weeks
Body weight | Change from Baseline at 12 weeks
Barriers to Insulin Treatment questionnaire | Change from Baseline at 12 weeks
  Measures aspects of psychological obstacles to insulin treatment in people with type 2 diabetes.
Diabetes Treatment Satisfaction Questionnaire | Change from Baseline at 12 weeks
  Designed to make the initial assessment of total diabetes treatment satisfaction, treatment satisfaction in specific areas, and perceived frequencies of hyperglycemia and hypoglycemia.
Short form 36 Health Survey | Change from Baseline at 12 weeks
  It is a generic measure, as opposed to disease specific, which assesses the relative burden of diseases, and differentiates the health benefits produced by a wide range of different treatments.
Adverse events | Collected throughout the study, average 14 weeks
Hypoglycemic events | Collected at baseline (on current insulin therapy) and throughout the study, average 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
No plan to share individual data sets, but will publish the results.

REFERENCES:
- [Derived] Mader JK, Lilly LC, Aberer F, Poettler T, Johns D, Trautmann M, Warner JL, Pieber TR. Improved glycaemic control and treatment satisfaction with a simple wearable 3-day insulin delivery device among people with Type 2 diabetes. Diabet Med. 2018 Oct;35(10):1448-1456. doi: 10.1111/dme.13708. Epub 2018 Jul 5. PMID 29888811